CLINICAL TRIAL: NCT03246711
Title: The Effect of 3rd Trimester Ramdan Fasting on Obestetric Outcome
Brief Title: Can Fasting Ramadan in the Third Trimester in Pregnancy Affects the Fetal Growth.
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, AYMAN ABDELKADER MOHAMED ABDELKADER, doctor, Ain Shams Maternity Hospital
Other Study IDs: AAMABDELKADER 2
Record Dates: First submitted 2017-07-22; First posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Fasting; Fetal Growth Retardation, Antenatal (Disorder)
MeSH Terms: conditions — Fasting; Fetal Growth Retardation | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Totally fasting: Fasting each day from sunrise to sunset the whole month
  Interventions: Behavioral: Fasting
- Partially fasting: means fasting from sunrise to sunset part of the month
  Interventions: Behavioral: Fasting
- Non fasting: women who did not fast at all

INTERVENTIONS:
Behavioral: Fasting — Totally or partially fasting the holy month of ramadan for muslims
  Groups: Partially fasting; Totally fasting

SUMMARY:
Prospective comparative cohort study including 159 pregnant women at the third trimester recruited from the antenatal clinic at EL-Demerdash outpatient clinic, and followed up during the holy month of Ramadan (from 18th June To 16th July 2015).

The patients recorded their pattern of fasting during Ramadan then grouped into three groups A, B, C regarding fasting state A- Non fasting group B- Partially fasting group C- Totally fasting group

.

DETAILED DESCRIPTION:
Many pregnant muslims women fast during Ramadan Since fasting during Ramadan is one of the five pillars of Islam and is a central part of Muslim culture, many women may fear a loss of connection with their communities or would feel guilty if they did not observe Ramadan. Each year, about 400 million out of 1 billion Muslims do this duty. Such tasks like eating, drinking, and smoking are forbidden from sunrise until sunset. Fasting during pregnancy has been always considered as a debatable condition.

Many women ask their obstetricians if fasting is safe for their baby or not? There have been many studies on metabolic changes and different aspects of human health during and after Ramadan .but there have been few studies on the effect of fasting on pregnancy outcome and there are also some controversies in the findings of different studies.

All mothers within the age range of 20 - 35 years and in the 3rd trimester pregnancy (starting from 28 weeks) which is going to be calculated according to the date of the last menstrual period & confirmed ultrasonically, normal healthy women with average body mass index (BMI) and Women included have no medical disorder.

Women who fulfilled the eligibility criteria were subjected an ultrasound fetal biometry every 2 weeks till delivery and assess fetal weight after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 - 35 years.
* Third trimester pregnancy (starting from 28 weeks) which is going to be calculated according to the date of the last menstrual period & confirmed by ultrasonography.
* Normal healthy women with average body mass index (BMI). Normal range (18.5 to 25).
* Women included have no medical disorder.

Exclusion Criteria:

* History of systemic disorder.
* Smoking narcotics or alcohol use.
* Have previous history of fetal loss.
* Multiple pregnancies.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Prospective comparative cohort study including 159 pregnant women at the third trimester recruited from the antenatal clinic at EL-Demerdash outpatient clinic, and followed up during the holy month of Ramadan (from 18th June To 16th July 2015).
  The patients recorded their pattern of fasting during Ramadan then grouped into three groups A, B, C regarding fasting state A- Non fasting group B- Partially fasting group C- Totally fasting group
Sampling Method: Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2015-06-18 (Actual); Primary Completion 2015-07-17 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Fetal growth | through study completion ( from 28 weeks pregnancy till delivery)
  assessment of the fetal growth biometry ( estimated fetal weight) every two weeks,

SECONDARY OUTCOMES:
neonatal weight | at the time of delivery of each participant
  measured in grams after delivery
mode of delivery | at the time of delivery of each participant
  percentages of emergency CS due to presumed fetal compromise

IPD SHARING:
Plan to Share IPD: Yes
no confidential data will be shared
Supporting Information: Study Protocol, CSR
Time Frame: december 2019

DOCUMENTS (2):
  • Study Protocol (2015-01-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT03246711/Prot_000.pdf
  • Statistical Analysis Plan (2015-10-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT03246711/SAP_001.pdf